NCT03545113 Unique Protocol ID: IRB00050577

Official Title: A randomized pilot study comparing graft-first to fistula-first strategies in older patients

with incident end-stage kidney disease

Date: 3/31/2020



## **Informed Consent Document**

**Project Title:** A randomized pilot study comparing graft-first to fistula-first strategies in older patients with incident end-stage kidney disease

Principal Investigator: Mariana Murea, M.D.

Co-Investigators: Jasmin Divers, Ph.D, Randolph Geary, M.D., Shahriar Moossavi M.D.,

Jennifer Gabbard, M.D., Isai Bowline, M.D.

## INTRODUCTION

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you have advanced Chronic Kidney Disease expected to require hemodialysis or End Stage Renal Disease, are undergoing hemodialysis, and your Kidney Doctor has determined that you need and are surgically eligible for permanent vascular access placement of a fistula or graft for your hemodialysis treatments. A vascular access is a surgically created vein or graft used to remove and return blood during hemodialysis. A fistula is a connection, made by a vascular surgeon, of an artery to a vein. A graft is a looped, plastic tube that connects an artery to a vein. When catheters are used for hemodialysis, it is best to be able to switch to using either a fistula or a graft. Catheters are considered temporary access because the goal is to be able to remove the catheter once there is a fistula or a graft that can be used for dialysis. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may





Picture source: Hemodialysis. What you need to know. National Kidney Foundation. www.kidney.org

# WHY IS THIS STUDY BEING DONE?

Many older adults require hemodialysis for advanced chronic kidney disease, but it is not clear which permanent vascular access method (fistula or graft) is best in terms of effectiveness and patient satisfaction. National guidelines require placement of a fistula or graft in patients on hemodialysis in order to experience better survival. The advantages of a fistula over a graft are not well known, especially in older population. Fistulas often fail to work after surgical placement and require repeated surgical interventions in order to be used for hemodialysis. Once a fistula develops, it may last for a longer period of time than a graft. Grafts have a higher chance to work and can be used sooner after placement. In this study, we will determine if placement of a graft access will be more effective at having your access switched from catheter to using the graft; have fewer interventions on the graft access; have better arm function; have better self-sufficiency with daily activities; and better quality of life compared to those who receive a fistula. We hope to identify strategies that decrease dialysis access failure and improve quality of life.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

Approximately eighty (80) people will take part in this pilot study.

#### WHAT IS INVOLVED IN THE STUDY?

If you agree to participate in this study by signing this consent form, you will be randomized to either have a graft or a fistula surgically placed in your arm. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance to be placed into either group. Patients randomized to receiving a graft will undergo surgical placement of a graft access in the forearm or arm by an experienced surgeon within 90 days of signing this consent form. Patients randomized to receiving a fistula will undergo surgical creation of a fistula access in the forearm or arm by an experienced surgeon within 90 days of signing this consent form.

Your Kidney Doctor has already determined that you need and are surgical eligible to undergo surgical intervention for either placement of a graft or creation of a fistula in order to be able to remove the catheter and use the new access for your future hemodialysis treatments. Your surgery will be done at Wake Forest Baptist Medical Center Medical Center Blvd. Winston-Salem, NC 27157 or any other Wake Forest affiliated institution (i.e., High Point Regional Medical Center).

The surgical intervention for placement of a graft or creation of a fistula will be done according to standard of care.

- The study staff, your kidney doctor, the surgeon and the anesthesiologist will explain to you the surgical procedure.
- The purpose of the surgery is to connect a large vein in the arm to a nearby artery, either directly (fistula surgery) or indirectly by inserting a graft material (graft surgery).
- You will receive regional anesthesia (numbing medicine) in your arm and medications for sedation. During regional anesthesia, a medicine is put through a needle or tube near nerves of your arm. You will temporarily lose feelings and movement of your arm. You will have pain relief for a period of time after surgery.
- Intubation (being put on a breathing machine) or blood transfusion is rarely required.
- After the procedure, you may be prescribed pain medication if needed.
- After the surgery, you will be monitored for a few hours and if your medical status is stable, you will be able to go home.

You will receive medical care after placement of graft or fistula according to standard care and as directed by your kidney doctor and/or primary care doctor. After this surgery, the evaluation for the function of either the graft or fistula will follow according to usual clinical practice. You will be examined in the medical office or at your dialysis unit on a regular basis by your kidney doctor, physician assistant, and nurses experienced in the care of grafts and fistulas. Any abnormalities that relate to either the graft or the fistula (such as changes on how the access looks or feels) will be addressed as directed by your kidney doctor. Interventions that may be needed for the graft or for the fistula after the surgery will be done according to your kidney doctor or surgeon's recommendations.

There will not be any changes in your usual medical care if you participate.

All of the following evaluation and reports will be performed and gathered specifically for this study at your dialysis session or at your regular doctor office visit by our study personnel.

- You will be asked to provide information from your health record such as age, sex, ethnic background, medical history, current medications, diet, exercise and medical care.
- You will be asked to complete a questionnaire (KDQOL-SF) to assess your health and how you are feeling, will be asked questions about your regular daily activities (ADL, IADL), and will be asked to perform a grip strength test at four to five different time points during your participation of the study.
- You will be asked questions about your satisfaction with the dialysis access (graft or fistula) (SF-VAQ) and about any pain in your graft or fistula (VDS or modified Abbey Pain Scale) at three to four different time points during your participation of the study.

- You will be asked to perform a timed 4 meter walk to test your walking speed.
- During the study you may be asked questions about your study participation experience.

There will be no medical visits and no blood collections done specifically or exclusively for this study. Information routinely gathered as part of your medical care will also be used in the study. Results of routine tests will be available to your doctor, and will be used to help determine study outcomes.

We can send copies of your test results to your primary doctor. Even if you do not wish to have any of your medical information sent to your physician, you can still participate in this research study.

Do you request that we send important medical findings from your study tests/exams to your personal physician?

| Γ. | Yes | [ ] No | Initials |
|----|--------|----------|------------|
| | 1 - 00 | 1 1 1 10 | 1111111111 |

## HOW LONG WILL I BE IN THE STUDY?

Your participation in this study will be for about 6 months. After the 6-month period, no study specific assessments/questionnaires will be performed, but we will continue to collect medical information from the medical records for approximately 3 years. You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. Your medical care will not be affected by your decision.

#### WHAT ARE THE RISKS OF THE STUDY?

Being in this study may involve some risk to you. You should discuss the risk of being in this study with the study staff.

- There is a slight risk that other people outside the study may access your information. We will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.
- Risks associated with surgery for placing a graft.

# Common risks/side effects:

- bleeding, pain, swelling or fluid collection at incision site
- soreness, numbness or bruising at incision site from anesthesia
- unable to use the graft or fistula as expected after surgery and requirement of another procedure or another surgery.

# Uncommon risks/side effects:

- decreased blood flow to hand or nerve damage resulting in hand numbness

#### Rare risks/side effects:

- infection at the incision site
- rupture of a blood vessel
- allergic reaction related to medications administered during or after surgery
- medical risk of surgery, such as cardiac event (.e.g, heart attack), respiratory failure, cerebrovascular event (e.g., stroke)
- intubation (placing a tube in the wind pipe to help you breath)
- blood transfusion
- nerve injury (lingering numbness, decreased sensation or permanent weakness) of the arm from anesthesia (The overall risk of long-term nerve injury is around 0.2%)
- Risks associated with surgery for creating a fistula.

#### Common risks/side effects:

- pain, swelling or fluid collection at incision site
- soreness, numbness or bruising at incision site from anesthesia

## Uncommon risks/side effects:

- decreased blood flow to hand or nerve damage resulting in hand numbness

# Rare risks/side effects:

- rupture of a blood vessel
- allergic reaction related to medications administered during or after surgery

- lack of vascular access maturation and requirement of a subsequent procedure or another surgery
- infection at the incision site
- medical risk of surgery, such as cardiac event (.e.g, heart attack), respiratory failure, cerebrovascular event (e.g., stroke).
- intubation (placing a tube in the wind pipe to help you breath)
- blood transfusion
- nerve injury (lingering numbness, decreased sensation or permanent weakness) of the arm from anesthesia (The overall risk of long-term nerve injury is around 0.2%)

An important, although very rare, complication of the regional nerve blocks (regional anesthesia) for both the fistula and graft surgery, is the development of a pneumothorax (air trapped between the lung and the rib cage). In the unlikely case you do develop a pneumothorax, you may not notice any changes immediately but you might develop breathing symptoms like persistent coughing, chest pain, shortness of breath within 24 hours after performance of the block. If any of those symptoms occur you should contact your medical doctor or go to the nearest emergency room immediately. An x-ray will confirm the diagnosis of pneumothorax and sometimes the evacuation of the air with a chest tube is necessary. Because this is a rare but serious side effect, you should be aware of those symptoms.

An independent Safety Officer will be reviewing the data from this research throughout the study.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future.

Based on experience with the surgical placement of a graft in patients who require hemodialysis, researchers believe it may be as good as standard therapy you could receive without being in the study but with fewer side effects. Because individuals respond differently to therapy, no one can know in advance if it will be helpful in your particular case.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options: to have a fistula or

graft which are the only standard of care procedures. Fistulas often fail after surgical placement and require repeated surgical interventions in order to be used for hemodialysis. Once a fistula develops, it may last for a longer period of time than a graft. Grafts have a higher chance to work and can be used sooner after placement. Dialysis catheters are used only in cases where a fistula or graft cannot be placed. Dialysis catheters carry a very high risk of infections and mortality associated with infections.

#### WHAT ARE THE COSTS?

There are no costs to you for taking part in this study. Costs for your regular medical care will be your own responsibility.

# WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or bio specimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or bio specimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by the National Institute of Health (NIH) which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in

this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document. Your individual research test result will not be included in your medical records.

## WILL YOU BE PAID FOR PARTICIPATING?

You will be compensated \$50 after you complete all study related procedures.

## WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the National Institutes of Health.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call the study investigator **Dr. Mariana Murea**, **M.D. at** 

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes: date of birth, contact information (address, telephone number, etc.), past medical history, laboratory results, procedures, other test results, how you respond to study procedures, and information from questionnaires, assessments and physical examinations. If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study may be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board (IRB); representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS), The National Institutes of Health (NIH) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to your original medical record for verification of clinical trial procedures or data, without violating your confidentiality and to the extent permitted by other applicable laws.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health

Information is shared with any of these groups it might no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept indefinitely. This authorization does not expire. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Dr. Mariana Murea that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:

# Mariana Murea, M.D.

Associate Professor, Internal Medicine/Nephrology

However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

#### WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Mariana Murea, M.D. at after hours).

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at

You will be given a copy of this signed consent form.

#### **Signatures**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

Please read the following sentence and think about your choice. After reading the sentence, circle YES or NO. If you have questions, please talk to your doctor or nurse.

You agree that your Wake Forest Baptist Health electronic medical record may be accessed by designated study personnel for use in future research to learn about, detect, prevent, treat or cure other health problems. If you answer NO to this question, you may still participate in this study.

| YES NO | | |
|---|---|---|
| Subject Name (Printed) | | |
| Subject Signature | Date | Time AM / PM |
| Person Obtaining Consent (Printed) | | |
| Person Obtaining Consent (Signed) | Date | Time AM / PM |
| Legally Authorized Representative Name (Print) | : | |
| The above named Legally Authorized Represent subject based upon (specify health care power of | _ | |
| Relationship to the Subject: | | |
| Legal Representative Signature: Time: am / pm | | Date: |